CLINICAL TRIAL: NCT03122262
Title: WRHI 060 (ADVANCE): A Randomised, Phase 3 Non-inferiority Study of DTG + TAF + FTC Compared With DTG + TDF + FTC and EFV + TDF + FTC in Patients Infected With HIV-1 Starting First-line Antiretroviral Therapy - Extension to 192 Weeks
Brief Title: ADVANCE Study of DTG + TAF + FTC vs DTG + TDF + FTC and EFV + TDF+FTC in First-line Antiretroviral Therapy
Acronym: ADVANCE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Professor Francois Venter (Other)
Responsible Party: Sponsor-Investigator, Professor Francois Venter, Professor, University of Witwatersrand, South Africa
Organization: University of Witwatersrand, South Africa (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WRHI060
Record Dates: First submitted 2016-10-11; First posted 2017-04-20 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: HIV-1 Infection
Keywords: Antiretroviral Agents, first-line antiretroviral therapy; dolutegravir; Tenofovir alafenamide
MeSH Terms: interventions — dolutegravir; tenofovir alafenamide; emtricitabine tenofovir alafenamide; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Tablets; Efavirenz, Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Tenofovir Alafenamide (Active Comparator): Descovy: Tenofivir alafenamide tablets 25mg daily, Emtricitabine 200mg daily
  Interventions: Drug: Dolutegravir; Drug: Tenofovir Alafenamide
- Dolutegravir (Active Comparator): Dolutegravir 50mg daily, Truvada 500mg daily
  Interventions: Drug: Dolutegravir; Drug: Truvada
- Atripla (Active Comparator): Atripla: Efavirenz 600mg daily, Tenofovir Disoproxil Fumarate 300mg daily, Emtricitabine 200mg daily
  Interventions: Drug: Atripla

INTERVENTIONS:
Drug: Dolutegravir — DTG 50mg Oral Tablet once daily
  Other Names: Tivicay
  Arms: Dolutegravir; Tenofovir Alafenamide
Drug: Tenofovir Alafenamide — TAF/FTC 25/200mg Oral Tablet once daily
  Other Names: Descovy
  Arms: Tenofovir Alafenamide
Drug: Truvada
  Other Names: TDF/FTC 300/200mg Oral Tablet
  Arms: Dolutegravir
Drug: Atripla
  Other Names: EFV/TDF/FTC 600/200/300mg Oral Tablet
  Arms: Atripla

SUMMARY:
This is a non-inferiority (10% non-inferiority margin), study to assess the efficacy and safety of dolutegravir, DTG (50 mg once daily [QD]) administered in combination with tenofovir alafenamide fumarate, TAF (25 mg QD) and emtricitabine, FTC (200 mg QD) compared to DTG (50 mg QD) administered in combination with tenofovir disoproxil fumarate, TDF (300 mg QD) and FTC (200 mg QD) and compared to efavirenz, EFV (600 mg QD) administered in combination with TDF (300 mg QD) and FTC (200 mg QD) through 96 weeks in patients with HIV-1 starting first-line ART.

DETAILED DESCRIPTION:
This is an open label randomised, non-inferiority (10% non-inferiority margin), phase 3 study to assess the efficacy and safety of DTG (50 mg once daily [QD]) administered in combination with TAF (25 mg QD) and FTC (200 mg QD) compared to DTG (50 mg QD) administered in combination with TDF (300 mg QD) and FTC (200 mg QD) and compared to EFV (600 mg QD) administered in combination with TDF (300 mg QD) and FTC (200 mg QD) through 96 weeks in patients with HIV-1 starting first-line ART.

Approximately 1110 male and female patients infected with HIV-1 who are eligible for first-line ART will be randomly assigned in a 1:1:1 ratio (approximately 370 patients per treatment group) to Treatment Group 1 (DTG + TAF + FTC) or Treatment Group 2 (DTG + TDF + FTC) or Treatment Group 3 (EFV + TDF + FTC). To ensure adequate representation of adolescents (12 - 18 years) in any treatment group, randomisation will be stratified according to age greater or less than 18 years. The study includes screening and baseline visits, 8 study visits from Week 4 to Week 84, and a preliminary end of study visit at Week 96.

The study will then take patients on Treatment Group 1 (DTG + TAF + FTC) or Treatment Group 2 (DTG + TDF + FTC) or Treatment Group 3 (EFV + TDF + FTC), who have completed 96 weeks successfully, and follow them to 192 weeks, with visits every 24 weeks after enrolment to 192 weeks. Study medication pill counts will be performed at each follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 12 years and ≥ 40 kg
2. Documented laboratory diagnosis of infection with HIV-1 (positive enzyme-linked immunosorbent assay HIV-1 antibody test) at screening
3. Plasma HIV-1 RNA (VL) ≥ 500 copies/mL
4. All pre-existing medical or laboratory abnormalities must be deemed to be stable by the investigator prior to study enrolment
5. Calculated creatinine clearance (CrCl) > 60 mL/min (Cockcroft-Gault formula) in > 18 years old OR > 80 mL/min (modified Cockcroft-Gault) in ≤ 18 years old
6. Ability to comprehend the full nature and purpose of the study, in the opinion of the investigator, and to comply with the requirements of the entire study.

To enrol in extension post-96 weeks:

Each patient must meet all of the following criteria to be enrolled in this study:

1. Previously enrolled on the ADVANCE study, and followed to week 96 (including those on post-trial access)
2. Ability to comprehend the full nature and purpose of the study, including the extended timeline, in the opinion of the investigator, and to comply with the requirements of the entire study.

Exclusion Criteria:

1. Previously received more than 30 days of treatment with any form of antiretroviral therapy (ART) or
2. Received any antiretrovirals within the last 6 months
3. Women who are pregnant at the time of the screening or baseline visit
4. Active tuberculosis and/or are on antituberculous therapy at the time of the baseline visit
5. Taking and cannot discontinue prohibited concomitant medications listed in 7.3 at least 2 weeks prior to the baseline visit and for the duration of the study period
6. Clinically unstable, in the investigator's opinion
7. Current history of drug or alcohol abuse that, in the opinion of the investigator, may be an impediment to patient adherence to the protocol
8. Patients who participated in a study with an investigational drug within 60 days of screening or who are currently receiving treatment with any other investigational drug or device may be ineligible to participate. This is an investigator decision
9. Have a strong likelihood of relocating far enough to make access to the study site difficult
10. History or presence of allergy to the study drugs or their components
11. Unstable liver disease (as defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminaemia, oesophageal or gastric varices, or persistent jaundice), cirrhosis, known biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones); Child-Pugh C.

To enrol in extension post-96 weeks:

Patients meeting the following criteria will be excluded from the study:

1. HbA1c, lipids and blood pressures that are not responding to treatment, in the opinion of the investigator and in consultation with the principal investigator, justifying substitution of DTG or TAF
2. Clinically unstable, in the opinion of the investigator
3. Have a strong likelihood of relocating far enough to make access to the study site difficult.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1110 (Actual)
Dates: Start 2017-01-16 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-07-29 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with undetectable plasma HIV-1 RNA levels (< 50 copies/mL) at Week 48 | 48 weeks
  The proportion of participants with undetectable plasma HIV-1 RNA levels at Week 48, will be calculated for each treatment group and summarised.

SECONDARY OUTCOMES:
Proportion of patients with undetectable plasma HIV-1 RNA levels (< 50 copies/mL) at Week 48, 96, 144 and 192 | 192 weeks
  Using FDA snapshot algorithm
Proportion of patients with plasma HIV-1 RNA levels < 200 copies/mL at Week 192 | 192 weeks
  • Participants with undetectable plasma HIV-1 RNA levels will be defined as those with plasma RNA levels of < 200 copies/mL. Successes/responders will be defined as those participants on each regimen with undetectable plasma HIV-1 RNA levels at Week 192.
Time to virologic failure (defined as confirmed HIV-1 RNA levels ≥ 1000 copies/mL at week 12 - 24 or ≥ 200 copies/mL at or after week 24) | 24 weeks
  Time to virologic failure will be modelled by Cox regression.
Change from baseline in plasma HIV-1 RNA levels at each visit | At week 12, 24, 36, 60, 72, 84, 96, 120, 144, 168, 192
  Individual patient plasma HIV-1 RNA levels will be summarised and listed by treatment and visit, together with changes from screening/enrolment plasma HIV-1 RNA levels. Observations (linear and log transformed) will also be presented graphically, over time, in the form of line plots.
Change from baseline in plasma CD4 levels at each visit | At week 12, 24, 36, 60, 72, 84, 96, 120, 144, 168, 192
  Individual patient CD4 counts will be summarised and listed by treatment and visit, together with changes from screening/enrolment CD4 values. Observations (linear and log transformed) will also be presented graphically, over time, in the form of line plots.

OTHER OUTCOMES:
Nature and frequency of adverse events | Week 48, 96, 144, 192
  A summary table will be presented, summarised by treatment, SOC and preferred term including the number of patients dosed in treatment group and number and percentage of subjects with AEs.
Analysis of PK data in those developing TB | Over course of TB treatment in those developing TB, during 3 regular scheduled visits
  Participants in treatment groups 1 and 2 who develop TB during the study will have DTG trough levels (ng/mL) measured at routine scheduled three visits. Trough levels will also be measured in control subjects (without TB coinfection) in a 3:1 ratio.
Analysis of PK data in those becoming pregnant | Monthly
  Participants in treatment groups 1 and 2 who develop TB during the study will have DTG trough levels (ng/mL) measures will be measured in control non-pregnantsubjects in a 3:1 ratio.
Virological efficacy in the 12 - 18 year age group | Week 48, 96
  Proportion of patients with undetectable plasma HIV-1 RNA levels (< 50 copies/mL) at Week 48 and 96 in a subgroup analysis of this age-range

CONTACTS AND LOCATIONS:
Overall Officials: Willem Daniel Francois Venter, FCP (SA), Principal Investigator — Wits Reproductive Health & HIV Institute, University of the Witswatersrand
Locations (4):
- South Africa (4):
  - Shandukani Research Centre, Johannesburg, Gauteng
  - Charlotte Maxeke Johannesburg Academic Hospital, Johannesburg, Gauteng
  - Sunnyside Office Park, Johannesburg, Gauteng
  - Wits RHI Yeoville Clinic, Johannesburg, Gauteng

IPD SHARING:
Plan to Share IPD: Yes
The data that will be shared is all of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, ICF
Time Frame: Immediately following publication
Access Criteria: Anyone who wishes to access the data

REFERENCES:
- [Derived] Manne-Goehler J, Fabian J, Sokhela S, Akpomiemie G, Rahim N, Lalla-Edward ST, Brennan AT, Siedner MJ, Hill A, Venter WDF. Blood pressure increases are associated with weight gain and not antiretroviral regimen or kidney function: a secondary analysis from the ADVANCE trial in South Africa. J Int AIDS Soc. 2024 Jul;27(7):e26268. doi: 10.1002/jia2.26268. PMID 38978403
- [Derived] Cindi Z, Kawuma AN, Maartens G, Bradford Y, Sokhela S, Chandiwana N, Venter WDF, Wasmann RE, Denti P, Wiesner L, Ritchie MD, Haas DW, Sinxadi P. Pharmacogenetics of tenofovir clearance among Southern Africans living with HIV. Pharmacogenet Genomics. 2023 Jun 1;33(4):79-87. doi: 10.1097/FPC.0000000000000495. Epub 2023 Mar 6. PMID 37098852
- [Derived] Cindi Z, Maartens G, Bradford Y, Venter WDF, Sokhela S, Chandiwana NC, Haas DW, Sinxadi P. Genetic Associations with Weight Gain among South Africans who Initiated Dolutegravir-Containing and Tenofovir-Containing Regimens. J Acquir Immune Defic Syndr. 2021 Jul 1;87(3):1002-1009. doi: 10.1097/QAI.0000000000002661. PMID 33625064
- [Derived] Siedner MJ, Moorhouse MA, Simmons B, de Oliveira T, Lessells R, Giandhari J, Kemp SA, Chimukangara B, Akpomiemie G, Serenata CM, Venter WDF, Hill A, Gupta RK. Reduced efficacy of HIV-1 integrase inhibitors in patients with drug resistance mutations in reverse transcriptase. Nat Commun. 2020 Dec 1;11(1):5922. doi: 10.1038/s41467-020-19801-x. PMID 33262331
- [Derived] Venter WDF, Sokhela S, Simmons B, Moorhouse M, Fairlie L, Mashabane N, Serenata C, Akpomiemie G, Masenya M, Qavi A, Chandiwana N, McCann K, Norris S, Chersich M, Maartens G, Lalla-Edward S, Vos A, Clayden P, Abrams E, Arulappan N, Hill A. Dolutegravir with emtricitabine and tenofovir alafenamide or tenofovir disoproxil fumarate versus efavirenz, emtricitabine, and tenofovir disoproxil fumarate for initial treatment of HIV-1 infection (ADVANCE): week 96 results from a randomised, phase 3, non-inferiority trial. Lancet HIV. 2020 Oct;7(10):e666-e676. doi: 10.1016/S2352-3018(20)30241-1. PMID 33010240
- [Derived] Venter WDF, Moorhouse M, Sokhela S, Fairlie L, Mashabane N, Masenya M, Serenata C, Akpomiemie G, Qavi A, Chandiwana N, Norris S, Chersich M, Clayden P, Abrams E, Arulappan N, Vos A, McCann K, Simmons B, Hill A. Dolutegravir plus Two Different Prodrugs of Tenofovir to Treat HIV. N Engl J Med. 2019 Aug 29;381(9):803-815. doi: 10.1056/NEJMoa1902824. Epub 2019 Jul 24. PMID 31339677